CLINICAL TRIAL: NCT00723918
Title: NARC 011: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of Methadone and Combination of Methadone and SAB378 in HIV-associated Painful Peripheral Neuropathy
Brief Title: Combination of an Investigational Cannabinoid and Methadone for HIV-associated Neuropathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of pharmaceutical support from Novartis - no participants randomized
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01NS32228_NARC011; NARC 011; U01NS032228 (NIH)
Record Dates: First submitted 2008-07-28; First posted 2008-07-29 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: HIV-associated Neuropathy; Polyneuropathy
Keywords: HIV-associated neuropathy; HIV; AIDS; cannabinoid; Cannabis; methadone; distal sensory polyneuropathy; polyneuropathy
MeSH Terms: conditions — Polyneuropathies; Acquired Immunodeficiency Syndrome; Marijuana Abuse | interventions — nabiximols; Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): methadone plus SAB placebo
  Interventions: Drug: methadone; Drug: SAB placebo
- 2 (Experimental): methadone plus active SAB
  Interventions: Drug: SAB378; Drug: methadone
- 3 (Placebo Comparator): methadone placebo plus SAB placebo
  Interventions: Drug: SAB placebo; Drug: Methadone placebo

INTERVENTIONS:
Drug: SAB378 — SAB 15 mg per day for 5 days, the 15 mg BID (twice a day) for 5 days, then 15 mg TID (three times a day) to end of 28-day treatment period, in combination with active methadone 5 mg BID for 5 days, then 5 mg TID for 5 days, to maximum of 10 mg TID until end of 28-day treatment period
  Other Names: SAB
  Arms: 2
Drug: methadone — Methadone 5 mg BID (twice a day) for 5 days, then 5 mg TID (three times a day) for 5 days, to maximum of 10 mg TID, in combination with SAB placebo or SAB active drug titrated as above, to end of 28-day treatment period.
  Arms: 1; 2
Drug: SAB placebo — an inactive substance
  Arms: 1; 3
Drug: Methadone placebo — Methadone placebo
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effectiveness of methadone alone and in combination with SAB378 for the treatment of painful HIV-associated neuropathy.

DETAILED DESCRIPTION:
Distal sensory polyneuropathy is the most common neurological complication of HIV disease and its treatment. To date no standard effective therapy has been identified.

In this study, scientists will evaluate the effectiveness of treating HIV-associated neuropathy with methadone alone and in combination with a novel cannabinoid SAB378. A cannabinoid is a molecule found only in the Cannabis plant. Cannabis and some cannabinoids are effective analgesics or pain relievers. The rationale for combination therapy is twofold: (1) medications with unique mechanisms of action may affect different aspects of neuropathic pain and (2) combination therapy may act synergistically-meaning the combined effect may be greater than the effect of each drug alone.

Approximately 84 participants will be enrolled in this double-blind, placebo-controlled, crossover study. Participants will be randomly assigned to three treatment groups-those receiving methadone and SAB378 placebo (an inactive substance), those receiving methadone and active SAB378, or those receiving methadone placebo and SAB378 placebo. All participants will be exposed to each of the 3 treatment groups during the study.

This trial is part of the Neurologic AIDS Research Consortium, an effective collaborative clinical study group dedicated to the study of HIV-associated neurological disease.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* HIV-associated neuropathy diagnosed by a neurologist
* Presence of at least a moderate pain score on the basis of completion of a baseline pain diary
* Stable antiretroviral regimen for at least 8 weeks prior to study entry.
* Hemoglobin ≥ 8.0 g/dL for males and ≥ 7.5 g/dL for females

Exclusion Criteria:

* Active AIDS-defining opportunistic infection within 45 days prior to study entry
* Renal insufficiency
* Chronic liver disease
* B12 deficiency
* Family history of hereditary neuropathy
* Discontinuation of dideoxynucleoside NRTI within 16 weeks prior to entry
* On neuroregenerative therapy
* Treatment with neurotoxic drugs within 120 days prior to entry
* Respiratory compromise
* Hypotension
* Active substance abuse or dependence
* History of alcohol-related complications within 6 months prior to screening
* Women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of methadone alone versus methadone and SAB378 for treatment of HIV-associated neuropathy | At the end of each 4-week treatment period

SECONDARY OUTCOMES:
Effect on quality of life, emotional functioning, cognitive functioning, safety | At the end of each 4-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: David B. Clifford, MD, Principal Investigator — Professor of Neurology, Washington University
Locations (3):
- United States (3):
  - University of California, San Diego, San Diego, California
  - University of New York Downstate Medical Center, Brooklyn, New York
  - University of Rochester, Rochester, New York